CLINICAL TRIAL: NCT04735055
Title: Artificial Intelligence Application in Predicting Disease Severity in Acute Pancreatitis
Brief Title: Artificial Intelligence Prediction for the Severity of Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Ali Tüzün İnce, Principal investigator, Bezmialem Vakif University
Other Study IDs: MLKkrm986%
Record Dates: First submitted 2020-09-30; First posted 2021-02-02 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Acute Pancreatitis; Artificial Intelligence; Outcome, Fatal
Keywords: Acute pancreatitis, Artificial intelligence,
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Artificial intelligence (AI) machine learning group: 90% machine learning part has also been divided into 2 parts as 70% for AI learning and 30% for testing the learning.
  70% of the acute pancreatitis patients (approximately 840 pts) will form the model training group of the study. 30% of the acute pancreatitis patients (approximately 360 pts) will form the testing group of the study.
  Since cross-validation will also be applied to the model here, the data will also change within itself, and also the distribution will be optimized to increase the predictive power.
- Validation group: 10% of the acute pancreatitis patients (approximately 134) will form the validation group of the study.
  Since cross-validation will also be applied to the model here, the data will also change within itself, and also the distribution will be optimized to increase the predictive power.

SUMMARY:
The incidence of acute pancreatitis (AP) is increasing nowadays. The diagnosis of AP is defined according to Atlanta criteria with the presence of two of the following 3 findings; a) characteristic abdominal pain b) amylase and lipase values ≥3 times c) AP diagnosis in ultrasonography (USG), magnetic resonance imaging (MRI), or computerized tomography (CT) imaging. While 80% of the disease has a mild course, 20% is severe and requires intensive care treatment. Mortality varies between 10-25% in severe (severe) AP, while it is 1-3% in mild AP.

Scoring systems with clinical, laboratory, and radiological findings are used to evaluate the severity of the disease. Advanced age (>70yo), obesity (as body mass index (BMI, as kg/m2), cigarette and alcohol usage, blood urea nitrogen (BUN) ≥20 mg/dl, increased creatinine, C reactive protein level (CRP) >120mg/dl, decreased or increased Hct levels, ≥8 Balthazar score on abdominal CT implies serious AP. According to the revised Atlanta criteria, three types of severity are present in AP. Mild (no organ failure and no local complications), moderate (local complications such as pseudocyst, abscess, necrosis, vascular thrombosis) and/or transient systemic complications (less than 48h) and severe (long-lasting systemic complications (>48h); organ insufficiencies such as lung, heart, gastrointestinal and renal). Although Atlanta scoring is considered very popular today, it still seems to be in need of revision due to some deficiencies in the subjects of infected necrosis, non-pancreatic infection and non-pancreatic necrosis, and the dynamic nature of organ failure. Even though the presence of 30 severity scoring systems (the most accepted one is the APACHE 2 score among them), none of them can definitely predict which patient will have very severe disease and which patient will have a mild course has not been discovered yet.

Today, artificial intelligence (machine learning) applications are used in many subjects in medicine (such as diagnosis, surgeries, drug development, personalized treatments, gene editing skills). Studies on machine learning in determining the violence in AP have started to appear in the literature. The purpose of this study is to investigate whether the artificial intelligence (AI) application has a role in determining the disease severity in AP.

DETAILED DESCRIPTION:
In a retrospective way, 1550 patients who were followed up at the Gastroenterology Clinic of Bezmialem Foundation University between October 2010 and February 2020 period and who were diagnosed with AP according to Atlanta criteria were screened. After the removal of 216 patients with missing data, 1334 patients were included in the study for evaluation.

1. Patient demographic information; [age (yo), gender (male/female), cigarette/alcohol usage (as yes or no)], clinical information; [height (centimeters), weight (kilograms), BMI (as kg/m2), presence of diabetes mellitus and hypertension (yes or no)], etiology of AP such as gallstones, alcohol, etc., and laboratory tests those taken within the first 24 hours of the admission; [CRP level (mg/dl, normally: 0-5), BUN level (mg/dl, normally; 9,8 - 20,1), creatinine level (mg/dl, normally; 0,57 - 1,11), number of leukocytes (normally 4.5 to 11.0 ×109/L) and hematocrit level (%, normally: 35,5-48%)], as well as Balthazar tomographic scoring [0: normal, 1: an increase in pancreatic size, 2: inflammatory changes in pancreatic tissue and peripancreatic fatty tissue, 3: irregularly bordered, single fluid collection, 4: irregularly bordered 2 or more fluid collections, 5 to 10 different degrees of necrosis)], will be recorded in the excel file.
2. Revised Atlanta scoring will also be recorded within a week period of hospital admission as mild, moderate, and severe scores. Infected pancreatic necrosis and sepsis that developed during the course of acute pancreatitis will be accepted as severe acute pancreatitis due to the inadequacy of some issues in Atlanta scoring. The severity of the disease will be evaluated according to the Atlanta scores. And the results of the artificial intelligence study will be matched according to the results of Atlanta scoring.
3. Complications are classified as 0; none, 2; local complications: pseudocyst, abscess, necrosis, thrombosis, and mesenteric panniculitis, 3; systemic complications: lung, kidney, gastrointestinal and cardiovascular complications, 4; mixed serious complications/co-morbidity situations, 5: infectious and septic complications.
4. Additionally, invasive procedure requirements such as endoscopic ultrasonography (EUS), endoscopic retrograde cholangiopancreatography (ERCP) (as yes or no), length of hospital stay (less than 10 days or more than 11 days), intensive care unit requirement (present or not), number of future AP attacks (in duration after a month of hospital admission, as of one attack or more than one attack), and survival (death, alive) will also be recorded.

Machine Learning Algorithm is used: Gradient Boosted Ensemble Trees Trees. ("Greedy Function Approximation: A Gradient Boosting Machine" by Jerome H. Friedman (1999)). The dataset has been partitioned with a 90%-10% ratio. 10% is for validation and 90% is for AI machine learning. 90% machine learning part has also been divided into two parts as 70% for AI Learning and 30% for testing the learning. For this purpose, 5-fold stratified sampling has been used

Artificial Intelligence Methods of the Study

Features Used for AI Machine Learning:

1. Gender: M/F
2. Age: Continuous Value
3. Height (cm): Continuous Value
4. Weight (Kg): Continuous Value
5. BMI Groups: Group 1: ≤ 25 kg/m2; Group 2; 25-30 kg/m2; Group 3: >30,1 kg/m2
6. Cigarette: 0; No, 1; Yes
7. Alcohol: 0; No, 1; Yes
8. Diabetes mellitus: 0; No, 1; Yes
9. Hypertension: 0; No, 1; Yes
10. Etiology: 1; biliary, 2; Alcohol, 3; hypertriglyceridemia, 4; hypercalcemia, 5; drug, 6; congenital, 7; cryptogenic, 8; endoscopic retrograde cholangiography (ERCP), 9; oddy sphincter dysfunction (OSD), 10; malignity, 11; intra papillary mucinous neoplasia (IPMN), 12: primary sclerosing cholangiography (PSC) 13: autoimmune, 14: multiple etiology
11. Leucocyte number (WBC): N; 4,5-11x100
12. Hematocrit (Hct): N; %35,5-48
13. C reactive protein (CRP): N: 0-5 mg/dl
14. Blood urea nitrogen (BUN): N: 9,8-20,1 mg/dl
15. Creatinine (KREA): N: 0,57-1,11 mg/dl
16. Baltazar Scoring (BLTZR): 0; Normal P, 1; Increase in pancreatic size, 2; Inflammatory changes in pancreatic tissue and peripancreatic fatty tissue, 3; Irregularly bordered, single fluid collection, 4, Irregularly bordered 2 or more fluid collections, with various degrees of necrosis (ranging between 5 and 10)

In Artificial Intelligence, Decision Tree Models are widely used for supervised machine learning. They may depend on the Gini index, gain ratio/entropy, chi-square, regression, and so on. In AI they are preferred because they generate understandable rules for humans unlike other machine learning algorithms such as Artificial Neural Networks and Support Vector Machines. On the other hand, they are considered to be weak learners. That means they are highly affected by noise and outliers existing in the data set. In order to go around this handicap, models like Random Forest, Ensemble Trees, Gradient Boosting have been developed.

Random forest and Ensemble trees generate rules by applying a certain decision tree algorithm to the portions of the data set vertically and horizontally. This technique dramatically reduces the error occurring in learning. After learning processes are completed, they combine weak decision trees into a strong and bigger decision tree model. Ensemble learning models achieve better learning by minimizing the average value of the loss function on the training set via a F ̂(x) approximation. The idea is to apply a steepest descent step to the minimization problem in a greedy fashion.

In this study, the gradient boost tree model which was proposed by Friedman has been used for machine learning. This model chooses a separate optimal value for each of the tree's parts rather than a single one for the whole tree. This approach can be used to minimize any differentiable loss L(y, F) in conjunction with forwarding stage-wise additive modeling. It is reported that the gradient boosting tree model outperforms random forest and regular ensemble trees in many cases.

The goal of the algorithm is to find an approximation F_m (x_i) which minimizes the expected L(y,F(x)) loss function.

The algorithm may be summarized as follows:

Inputs:

A training data set: {(x_i,y_i )} i=1 to n with n dimension and a class variable A differentiable loss function: L(y,F(x)) The number of iterations: M.

Output:

F_m (x_i)

Algorithm:

Initialize the model with a constant value:

F_0 (x)=arg min⁡∑_(i=1)^n▒〖L(y_i,γ)〗

For m = 1 to M:

Compute pseudo-residuals rim r_im=-[(∂L(y_(i,) F(x_i )))/(∂F(x_i))]

Train a base learner to pseudo-residuals, using the training set:

{(x_i,y_i )} i=1 to n Compute multiplier γ γ=arg min⁡∑_(i=1)^n▒〖L(y_i,F_(m-1) (x_i )+γh_m (x_i ))〗

Update the model:

〖F_m (x_i)=F〗_(m-1) (x_i )+γ_m h_m (x_i ) Output F_m (x_i)

In the analysis, Synthetic Minority Oversampling Technique (SMOTE) [5] has been used in order to avoid the disadvantage of class variable imbalance. SMOTE is a data augmentation technique to increase data. In some cases, the class variable may not have an equal amount of values from all cases. For example, there may be much more survived patients than those who lost their lives. In this kind of situation, data are augmented. There was an imbalance in the class variables in the data set of this study. So, SMOTE has been applied to increase the minority classes for training.

The dataset has been partitioned with a 90%-10% ratio. 10% is for validation and 90% is for AI machine learning. 90% machine learning part has also been divided into two parts as 70% for AI Learning and 30% for testing the learning. For this purpose, 5-fold stratified sampling has been used. KNIME analytic platform has been used for the AI machine learning.

ELIGIBILITY:
Inclusion Criteria:

- Patients with acute pancreatitis diagnosis who admitted to ER within 24 hours after the beginning of abdominal pain

Exclusion Criteria:

* Patients who sign a treatment rejection form immediately after admission to the hospital and leave the hospital
* Patients with uncompleted data
* Psychiatric patients
* Patients with very poor general conditions

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute pancreatitis diagnosis according to the Atlanta criteria
Sampling Method: Non-Probability Sample
Enrollment: 1334 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Accurately estimation of the severity of the disease by machine learning method | Within a week.
  Severity is described as mild, moderate, and severe acute pancreatitis according to the revised Atlanta criteria.

SECONDARY OUTCOMES:
Invasive procedure requirement | Within a week
  Need for EUS or ERCP during hospital stay for evaluation of the reasons such as distal choledochal obstruction by stone, pseudocyst or necrosis developments (As yes or no)
Intensive care unit requirement | Within a week
  Transferring the patient to the ICU where life support is needed in order to survive if patients have dyspnea (if respiratory rate is more than 25/minute), hypotension (less than 90/60 mmHg), if patient have gastrointestinal bleeding (more than 2 lt. in a day), if the patient's BUN level is higher than 20 mg's and progressively increases (as yes or no)
Survival status | Within a week
  Death: if patient is alive (yes) if dies (no)
Length of hospital stay | Within a month
  Durations lasted in hospital as a day (as less than 10 days or more than 10 days)
Number of AP attacks | After a month of hospital admission as one attack or more than one attack
  Admission to the hospital again with the AP attack.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Silahtaroğlu, Prof., Principal Investigator — Medipol University
Locations (1):
- Bezmialem Vakif University, Gastroenterology Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Fei Y, Gao K, Li WQ. Artificial neural network algorithm model as powerful tool to predict acute lung injury following to severe acute pancreatitis. Pancreatology. 2018 Dec;18(8):892-899. doi: 10.1016/j.pan.2018.09.007. Epub 2018 Sep 26. PMID 30268673
- [Background] van den Heever M, Mittal A, Haydock M, Windsor J. The use of intelligent database systems in acute pancreatitis--a systematic review. Pancreatology. 2014 Jan-Feb;14(1):9-16. doi: 10.1016/j.pan.2013.11.010. Epub 2013 Dec 4. PMID 24555973
- [Background] Yoldas O, Koc M, Karakose N, Kilic M, Tez M. Prediction of clinical outcomes using artificial neural networks for patients with acute biliary pancreatitis. Pancreas. 2008 Jan;36(1):90-2. doi: 10.1097/MPA.0b013e31812e964b. No abstract available. PMID 18192888
- [Background] Pearce CB, Gunn SR, Ahmed A, Johnson CD. Machine learning can improve prediction of severity in acute pancreatitis using admission values of APACHE II score and C-reactive protein. Pancreatology. 2006;6(1-2):123-31. doi: 10.1159/000090032. Epub 2005 Dec 1. PMID 16327290
- [Background] Andersson B, Andersson R, Ohlsson M, Nilsson J. Prediction of severe acute pancreatitis at admission to hospital using artificial neural networks. Pancreatology. 2011;11(3):328-35. doi: 10.1159/000327903. Epub 2011 Jul 9. PMID 21757970
- [Background] Qiu Q, Nian YJ, Guo Y, Tang L, Lu N, Wen LZ, Wang B, Chen DF, Liu KJ. Development and validation of three machine-learning models for predicting multiple organ failure in moderately severe and severe acute pancreatitis. BMC Gastroenterol. 2019 Jul 4;19(1):118. doi: 10.1186/s12876-019-1016-y. PMID 31272385
- [Background] Greedy function approximation: A gradient boostingmachine.
- [Background] Clustering, A. (2009). Clustering Categorical Data Using Hierarchies. Engineering and Technology, 1(2), 334-339.
- [Background] Silahtaroğlu, G. (2009). An Attribute-Centre Based Decision Tree Classification Algorithm. Engineering and Technology, 302-306.
- [Background] Bentéjac, C., Csörgő, A., & Martínez-Muñoz, G. (2021). A comparative analysis of gradient boosting algorithms. Artificial Intelligence Review, 54(3). https://doi.org/10.1007/s10462-020-09896-5.
- [Background] Bentéjac, C., Csörgő, A., & Martínez-Muñoz, G. (2021). A comparative analysis of gradient boosting algorithms. Artificial Intelligence Review, 54(3). https://doi.org/10.1007/s10462-020-09896-5
- [Background] Berthold, M. R., Cebron, N., Dill, F., Gabriel, T. R., Kötter, T., Meinl, T., … Wiswedel, B. (2009). KNIME - the Konstanz information miner. ACM SIGKDD Explorations Newsletter. https://doi.org/10.1145/1656274.1656280